CLINICAL TRIAL: NCT01374724
Title: Preventing Relapse Following Involuntary Smoking Abstinence
Acronym: AFV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Tennessee (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Minnesota (Other); United States Air Force (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: FWH20100149H-2; 1R01HL095785-01A1 (NIH)
Record Dates: First submitted 2011-06-14; First posted 2011-06-16 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2015-11

CONDITIONS: Smoking; Smoking Cessation
Keywords: Tobacco Use; Relapse Prevention; Military; Smokeless Tobacco Use; Dual Use
MeSH Terms: conditions — Smoking; Smoking Cessation; Tobacco Use | interventions — Secondary Prevention; Crisis Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ban & Informational Pamphlet (Experimental): Following 8.5 weeks of cessation subjects are given an informational pamphlet on tobacco cessation and relapse prevention.
  Interventions: Behavioral: Tobacco Use Ban; Behavioral: Informational Pamphlet
- Ban & Tailored Pamphlet (Experimental): After 8.5 weeks of tobacco use cessation during Basic Military Training subjects are provided a tailored relapse prevention pamphlet inspired by Forever Free and tailored for use in the United States Air Force
  Interventions: Behavioral: Tobacco Use Ban; Behavioral: Tailored Pamphlet
- Ban & Tailored Pamphlet & Intervention (Experimental): After 8.5 weeks of tobacco use cessation during Basic Military Training subjects are provided a tailored relapse prevention pamphlet inspired by Forever Free and tailored for use in the United States Air Force. In addition they are given a face to face relapse prevention intervention.
  Interventions: Behavioral: Tobacco Use Ban; Behavioral: Tailored Pamphlet; Behavioral: Relapse Prevention Intervention

INTERVENTIONS:
Behavioral: Tobacco Use Ban — Airmen are restricted from use tobacco products during Basic Military Training which lasts for 8.5 weeks.
  Other Names: Tobacco Ban
Behavioral: Tailored Pamphlet — A tailored relapse prevention pamphlet inspired by Forever Free and tailored for use in the United States Air Force.
  Other Names: Tailored tobacco cessation information
  Arms: Ban & Tailored Pamphlet; Ban & Tailored Pamphlet & Intervention
Behavioral: Informational Pamphlet — The National Cancer Institute Pamphlet "Clearing the Air" was provided to subjects.
  Other Names: Tobacco cessation pamphlets
  Arms: Ban & Informational Pamphlet
Behavioral: Relapse Prevention Intervention — A 15 - 30 minute relapse prevention intervention designed to increase motivation to remain tobacco free.
  Other Names: Relapse prevention; Motivational interventions; Brief interventions
  Arms: Ban & Tailored Pamphlet & Intervention

SUMMARY:
The prevalence of tobacco use in the military is too high. This study is designed to take advantage of the 8.5 weeks of forced tobacco cessation during Basic Military Training and develop effective interventions to prevent tobacco relapse.

Hypotheses or Research Questions:

* Are there differences in the rate of relapse between three groups participating in a tobacco abstinence maintenance intervention?
* Do the tobacco abstinence maintenance interventions delay relapse?

DETAILED DESCRIPTION:
Consented subjects will be randomly assigned either to:(a) National Cancer Institute tobacco cessation pamphlet , to (b) Tailored relapse prevention pamphlet , or to (c) Tailored relapse prevention pamphlet + 1 proactive relapse prevention face-to-face meeting.

To determine the long-term (12 month) efficacy of the abstinence maintenance intervention. Our primary outcome is abstinence from tobacco products at the 12 month follow-up. A secondary outcome will be to determine if these interventions delay relapse among those who relapse to smoking or other tobacco use.

Significance: Cigarette smoking use is the number one preventable cause of morbidity and mortality in this nation (CDC, 1999; Mokdad et al., 2004). Preventing relapse is a high priority for those attempting to quit smoking as most people who attempt cessation relapse within a very short period of time (Fiore et al., 2000). Of smokers who receive a formal cessation program, at least 70% relapse (Fiore et al., 2000); among self quitters, the relapse rate is approximately 90% (Cohen et al., 1989). It is still the case, however, that the vast majority of smokers who try to stop smoking do so with no or with minimal assistance (Garvey et al., 1992).

While the vast majority of smokers try to quit on their own, surprisingly little research has been conducted on reducing relapse among self-quitters. Brandon and colleagues (2000, 2003, 2004) have demonstrated that a series of 8 self-help printed materials consistently produced higher point-prevalence abstinence rates in smokers that had quit on their own. Given the enormous public health implications of this approach, more research on promoting long-term self-quitting is clearly needed. In addition a number of never smokers actually start smoking shortly after accession into the Air Force (Klesges et. al., 1999; 2006). The goal of this research is to encourage all airmen to remain tobacco free. Because of this the investigators are encouraging all airmen to participate in the abstinence maintenance interventions.

Military Relevance: Virtually all research to date on promoting self-quitting has been conducted in samples where participants have voluntarily stopped smoking prior to participating in the interventions (Brandon et al., 2000, 2004). However, nothing is known about methods of preventing and delaying initiation following involuntary abstinence (e.g., military training, during hospital stays, in jails, prisons, & psychiatric facilities). Previous research (Klesges et al., 1999, 2006) has determined that protracted involuntary cessation in the military with no other intervention is associated with significant long-term cessation rates (15-20% at a one-year follow-up). To our knowledge, no study has successfully intervened to reduce relapse rates following a protracted involuntary abstinence (such as in Basic Military Training).

ELIGIBILITY:
Inclusion Criteria:

* Active duty Air Force personnel
* Has smoked five or more cigarettes per day for at least 1 year before study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23000 (Estimated)
Dates: Start 2011-05; Primary Completion 2017-04 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Smoking cessation maintenance | 12 month follow-up
  Subjects will be called at one year post intervention to determine self-report of tobacco use status.

SECONDARY OUTCOMES:
Delayed relapse among those who relapse to tobacco use | 12 month follow-up
  Subjects will be contacted 12 months after the intervention to determine via self-report when they relapsed.

CONTACTS AND LOCATIONS:
Overall Officials: Robert C. Klesges, Ph.D., Principal Investigator — University of Tennessee Health Science Center and St. Jude Childrens' Research Hospital; Harry Lando, Ph.D., Principal Investigator — University of Minnesota; Gerald W. Talcott, Ph.D., Principal Investigator — University of Tennessee
Locations (2):
- United States (2):
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas

REFERENCES:
- [Derived] Brandon TH, Klesges RC, Ebbert JO, Talcott GW, Thomas F, Leroy K, Richey PA, Colvin L. Preventing smoking initiation or relapse following 8.5 weeks of involuntary smoking abstinence in basic military training: trial design, interventions, and baseline data. Contemp Clin Trials. 2014 May;38(1):28-36. doi: 10.1016/j.cct.2014.03.001. Epub 2014 Mar 15. PMID 24637237